CLINICAL TRIAL: NCT04004013
Title: A Randomised, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Effect of Lifenol in Improving Bone Status in Postmenopausal Osteopenic Women
Brief Title: Evaluate the Effect of Lifenol in Improving Bone Status in Postmenopausal Osteopenic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Givaudan France Naturals (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AFCRO-100
Record Dates: First submitted 2019-06-10; First posted 2019-07-01 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Osteopenia, Generalized
Keywords: osteopenia; phytoestrogen; hop; menopause
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifenol (Active Comparator): 50 participants who meet the eligibility criteria will be randomised under active arm and will receive Lifenol product during 12 months
  Interventions: Dietary Supplement: Lifenol®
- Placebo (Placebo Comparator): 50 participants who meet the eligibility criteria will be randomised under Placebo arm and will receive placebo product during 12 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lifenol® — Lifenol®, powdered extract obtained from female hops flowers (Humulus lupulus L.) standardized in 8-PN content (100 µg /day) + maltodextrin = 500 mg/capsule
  + 1000 mg of calcium and 800 IU of vitamin D per day
  Arms: Lifenol
Dietary Supplement: Placebo — Maltodextrin = 500 mg/capsule
  + 1000 mg of calcium and 800 IU of vitamin D per day
  Arms: Placebo

SUMMARY:
A Randomised, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Effect of Lifenol® in Improving Bone Status in Postmenopausal Osteopenic Women. 100 postmenopausal women will be enrolled to investigate the effect of a 12 month supplementation with Lifenol® on bone density DXA parameters and plasma bone biomarkers.

DETAILED DESCRIPTION:
Osteoporosis is a skeletal disorder characterized by reduced bone mass and deterioration in bone architecture leading to an increased bone fragility and fracture risk. Postmenopausal women are a particularly at-risk population as the maintenance of bone homeostasis is influenced by estrogens. Recently, phytoestrogens have drawn attention as an interesting natural way to prevent oestrogen-deficient osteoporosis. Hops contain one of the most potent phytoestrogen known to date: 8-prenylnaringenin (8-PN). Lifenol® is a polyphenolic powdered extract obtained by a patented process from the female hop flowers (Humulus lupulus L.), standardized in 8-PN content.

Therefore, the present clinical trial aims to determine whether long-term consumption of Lifenol® can reduce bone mineral density loss in postmenopausal women with osteopenia taking traditional recommended calcium and vitamin D supplementation (1000 mg of calcium and 800 IU of vitamin D per day).

100 postmenopausal women (>1 year post-menopause) will be enrolled to consume during 12 months either Lifenol® (dose of 100µg of 8-PN per day) or a placebo. Effect of investigational product will be measured notably on bone density DXA parameters and plasma bone biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent;
2. Be 50 - 85 years of age;
3. Be a free-living postmenopausal (> 1 year post menopause) woman;
4. Have a Body Mass Index (BMI) 18 - 32.0 kg/m²;
5. Present with a stable weight (+/- 3 kg) for at least the last three (3) months;
6. Be a non-smoker
7. Maintain existing food and physical activity patterns throughout the study period;
8. Present with osteopenia defined as a dual energy X-ray absorptiometry (DXA) T score comprised between -1 and -2.5;
9. Be willing to consume the investigational product daily for the duration of the study.

Be able to give written

Exclusion Criteria:

1. Are hypersensitive to any of the components of the investigational product;
2. Is currently involved in any other clinical trial or having participated in a trial within the preceding 60 days;
3. Has a diagnosis of osteoporosis (defined as a T score strictly inferior to -2.5);
4. Is currently a smoker;
5. Trying to lose weight for the last three (3) months (following a diet or exercise regimen designed for weight loss);
6. Recent (within 4 weeks) gastroenteritis or food borne illness;
7. Having taken antibiotics or laxatives during the preceding 2 months or anticipated consumption;
8. Currently taking (and during the past 3 months) any drug for osteoporosis (bisphosphonates, parathyroid hormone, strontium ranelate or denosumab);
9. Currently taking (and during the past 3 months) treatment with oestrogen or hormone therapy;
10. Currently taking (and during the past 3 months) treatment with oestrogen agonist or antagonist products (raloxifene or tamoxifene);
11. Currently taking any supplementation with isoflavones or foods fortified with isoflavones;
12. Currently taking (and during the past 4 weeks) any vitamin K supplementation.
13. Exhibiting excess alcohol consumption, defined as greater than 11 standard drinks per week for women or drug dependence,
14. Has a significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would preclude supplement ingestion and/or assessment of safety and the study objectives;
15. Has a known organic disease, including an inflammatory bowel disease, a benign or malign tumour of intestine or colon and significant systemic disease;
16. Has a history of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, or carcinoma in situ with no significant progression over the past 2 years;
17. Has uncontrolled hypertension (systolic or diastolic blood pressure superior to 160 and 110 respectively). Subject on hypertension medication, must be on stable medication for 3 months;
18. Has uncontrolled hypothyroidism or hyperthyroidism; subject must be stable on medication for 3 months
19. Current illnesses which could interfere with the study (e.g. prolonged severe diarrhoea, regurgitation/severe, difficulty swallowing).
20. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Bone mineral density at the L2-L4 lumbar spine region | baseline and 12 months
  Change of bone mineral density at L2-L4 lumbar spine region over 12 months.

SECONDARY OUTCOMES:
Bone mineral density at the femoral neck region | baseline, 6 and 12 months
  DXA scan will provide this parameter
Bone mineral content at the L2-4 lumbar spine and femoral neck region | baseline, 6 and 12 months
  DXA scan will provide this parameter
T-score | baseline, 6 and 12 months
  DXA scan will provide this parameter
Fracture risk assessment tool (FRAX) score | baseline, 6 and 12 months
  FRAX score will be calculated an online tool (university of sheffield frax tool).
Plasma bone biomarkers | baseline, 6 and 12 months
  Change in plasma bone biomarkers will be measured.
Plasma prenylflavonoids | baseline, 6 and 12 months
  Change in plasma prenylflavonoids will be measured.
Glucose homeostasis and lipid profile | baseline, 6 and 12 months
  Change in plasma glucose, insulin and lipids will be measured.
Quality of life evaluation | baseline, 3, 6, 9 and 12 months
  36-item short form (SF-36) will be performed to assess by quality of life.
Gastrointestinal tolerance evaluation | baseline, 3, 6, 9 and 12 months
  Gastrointestinal tolerance of the product will be assessed by the Gastrointestinal Symptom Rating Scale (GSRS).

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided
To revisit this after investigation period